CLINICAL TRIAL: NCT02418247
Title: Phase Ⅱ Non-randomized Multicenter Controlled Trial About Effect of Remnant Ablation Therapy on the Recurrence in Low-risk Differentiated Thyroid Cancer Patients
Brief Title: Minimize Radioactive Iodine Ablation Of Remnant Thyroid in Differentiated Thyroid Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Eun Kyung Lee, M.D., Ph.D., National Cancer Center, Korea
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS13-671; 1410650-1,2 (Other Grant/Funding Number: NCC Research Fund)
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Thyroid Neoplasms
Keywords: radioactive iodine therapy; ablation; thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Iodine-131; Iodine-123

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low dose RAI (Active Comparator): Low dose RAI (radioactive iodine I-131, 30mCi) will be given to ablate remnant thyroid tissue.
  Interventions: Drug: I131
- diagnostic RAI (Sham Comparator): Diagnostic RAI (radioactive iodine I-123, 2-6mCi) will be given to achieve postRAI scan.
  Interventions: Drug: I123

INTERVENTIONS:
Drug: I131
  Other Names: low dose RAI
  Arms: low dose RAI
Drug: I123
  Other Names: diagnostic RAI
  Arms: diagnostic RAI

SUMMARY:
The researchers investigated the rate of biochemical remission in patients without radioactive iodine therapy compared to patients with low dose radioactive iodine treatment in differentiated thyroid cancer patients who underwent total thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients with differentiated thyroid cancer
* recently underwent total thyroidectomy (within 6 months)
* pathological criteria

  1. T1bN0 : Tumor size 1-2cm with no microscopic extension with multifocality (within three foci)
  2. T3N0 : Tumor size <=2cm with microscopic extension (less than strap muscle)
  3. T1-3N1a : 3 or less micrometastatic lymph node

Exclusion Criteria:

* differentiated thyroid cancer with aggressive variant, poorly differentiated thyroid cancer, medullary thyroid cancer, anaplastic thyroid cancer
* gross extension (strap muscle or more)
* thyroid cancer with distant metastasis
* previous remote history of thyroid cancer surgery
* history of cervical external beam radiation therapy
* previous history of comorbid cancer within 5 years
* renal insufficiency (Ccr <30ml/min)
* women with pregnancy or breast feeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical Remission Rate | within 1 year since first thyroid hormone withdrawal regardless of radioactive iodine administration

CONTACTS AND LOCATIONS:
Overall Officials: Eun Kyung Lee, M.D.,Ph.D., Study Chair — National Cancer Center, Korea
Locations (5):
- South Korea (5):
  - Chungnam National University Hospital, Daejun
  - National Cancer Center, Korea, Goyang
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul National University Bundang Hospital, Sungnam